CLINICAL TRIAL: NCT03430440
Title: Comparison of Analgesic Effects According to Patient-controlled Epidural Analgesia Modes in Patients Undergoing Open Gastrectomy: a Randomized Controlled Trial
Brief Title: Comparison of Analgesic Effects According to Patient-controlled Epidural Analgesia Modes in Patients Undergoing Open Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2016-1152
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Open Gastrectomy With Gastric Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIPKA mode (Experimental): The newly developed computer-integrated patient-controlled analgesia (CIPCA) mode increases or decreases the basal infusion rate with the use of the patient's bolus button.
  Interventions: Device: Apply CIPKA mode
- Conventional mode (Active Comparator): The conventional mode in which only the basal infusion rate is set to be fixed.
  Interventions: Device: Conventional mode

INTERVENTIONS:
Device: Apply CIPKA mode — The newly developed computer-integrated patient-controlled analgesia (CIPCA) mode increases or decreases the basal infusion rate with the use of the patient's bolus button. Compared with the conventional mode in which only the basal infusion rate is set to be fixed, the CIPCA mode sets the basal infusion rate, the increase / decrease rate of basal rate, and the increment / decrement interval.
  Arms: CIPKA mode
Device: Conventional mode — PCA pumps typically set a fixed basal infusion rate to set the analgesic to enter at a constant rate every hour (conventional mode).
  Arms: Conventional mode

SUMMARY:
Epidural PCA (patient controlled analgesia) for post-operative pain management are effective analgesic method. It is widely used in the postoperative pain management for decades.

PCA pumps typically set a fixed basal infusion rate to infuse the analgesics at a constant rate per every hour (conventional mode). In contrast, the newly developed computer-integrated patient-controlled analgesia (CIPCA) mode increases or decreases the basal infusion rate with the use of the patient's bolus button. The CIPCA mode sets the basal infusion rate, the increase / decrease rate of basal rate, and the increment / decrement interval. If the patient presses the bolus button within the set time interval, the set infusion rate is increased because the analgesic is more required. If the bolus button is not pressed during the set time interval, the infusion rate is decreased. Therefore, it can be said that it is an effective method to control the dose of analgesic agent more sensitively to changes in patient's needs and pain.

ELIGIBILITY:
Inclusion Criteria:

1. elective open gastrectomy due to stomach cancer
2. ASA classification Ⅰ-Ⅲ

Exclusion Criteria:

1. hematologic clotting defect
2. sepsis
3. distance metastasis
4. PCA drug (fentanyl, Ropivacaine) allergy
5. Patients who can not read the consent form or are not fluent in Korean (illiterate, foreigner)
6. pregnant, lactating women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-11-11 (Estimated); Study Completion 2020-11-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain (numerical rating scale: 0 ~ 10) | at 6 hours postoperatively

SECONDARY OUTCOMES:
Postoperative pain (numerical rating scale: 0 ~ 10) | at 1, 24, and 48 hours after surgery
PCA total dose/additional analgesic dose | at 1, 6, 24, 48 hours after surgery
Side effects of PCA (area and vomiting / hypotension / muscle weakness | at 1, 6, 24, 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No